CLINICAL TRIAL: NCT00580060
Title: Injection Of AJCC Stage IIB, IIC, III And IV Melanoma Patients With A Multi-Epitope Peptide Vaccine Using GM-CSF DNA As An Adjuvant: A Pilot Trial To Assess Safety And Immunity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Miguel-Angel Perales, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-142; NCI Protocol #: 5906; NCT00085137 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Melanoma
Keywords: AJCC; stage; IIB; IIC; III; IV; Melanoma; HLA-A2+; Vaccine
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: GM-CSF DNA, NSC 683472 gp100: 209-217(210M), NSC 699048 Tyrosinase: 368-376(370D) — In the Dose Ranging part of the study, cohorts of 3 patients will be treated at increasing dose levels of GM-CSF DNA delivered subcutaneously (100, 400, or 800 mg), followed by administration of both peptides subcutaneously to the same site on day 5 or day 6. Patients will be treated monthly for three immunizations.
  Other Names: GM-CSF DNA; NSC 683472 gp100: 209-217(210M); NSC 699048 Tyrosinase: 368-376(370D)

SUMMARY:
This is a pilot trial to investigate the use of GM-CSF DNA as an adjuvant for peptide vaccination in patients with metastatic melanoma. The objective of this study is to determine the safety and adjuvant effect of vaccination with the gene coding for human GM-CSF with a multi-epitope melanoma peptide vaccine (tyrosinase and gp100 peptides) in patients with AJCC stage IIB, IIC, III and IV melanoma who are HLA-A2+. We will assess whether use of GM-CSF DNA is safe and generates an immune response to peptides derived from antigens on melanoma cells.

DETAILED DESCRIPTION:
This is a pilot trial to investigate the use of GM-CSF DNA as an adjuvant for peptide vaccination in patients with metastatic melanoma. The objective of this study is to determine the safety and adjuvant effect of vaccination with the gene coding for human GM-CSF with a multi-epitope melanoma peptide vaccine (tyrosinase and gp100 peptides) in patients with AJCC stage IIB, IIC, III and IV melanoma who are HLA-A2+. We will assess whether use of GM-CSF DNA is safe and generates an immune response to peptides derived from antigens on melanoma cells.

In the Dose Ranging part of the study, cohorts of 3 patients will be treated at increasing dose levels of GM-CSF DNA delivered subcutaneously (100, 400, or 800 ug), followed by administration of both peptides subcutaneously to the same site on day 5 or day 6. Patients will be treated monthly for three immunizations. Pharmacokinetic studies will be performed during the first cycle. Patients' peripheral blood mononuclear cells will be collected in order to measure the T cell responses induced by the vaccines. Toxicity will be assessed during this part of the study, although we do not expect to achieve a dose limiting toxicity (DLT). The dose for the second part of the study will be the maximum tolerated dose.

The second part of the study will assess the immunological efficacy of the vaccine. Nine patients will receive GM-CSF DNA delivered subcutaneously at one site, followed by administration of both peptides to the same site on day 5 or day 6, every month for three immunizations. A total of at least 18 patients is planned for both phases of the study. Patients' peripheral blood mononuclear cells will be collected in order to measure the T cell responses induced by the vaccines. Specifically, Elispot assays for CD8+ T cells responses against the peptides will be assessed, and will be the primary method to determine the generation of a specific immune response to the peptide antigens.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented malignant melanoma, American Joint Commission on Cancer (AJCC) stage IIB, IIC, III or IV (54). Patients with resectable stage IIB, IIC and III disease must have undergone surgical resection before participating in this study.
* Patients with choroidal melanoma may participate if they fulfill one of the following criteria: Basal diameter > or = 16 mm; Height > or = 8 mm or involvement of ciliary body with tumor.
* For all patients, pathology slides must be reviewed by the Pathology Department of Memorial Sloan-Kettering Cancer Center for confirmation of melanoma diagnosis.
* Patients must be HLA-A2 positive.
* Patients must weigh at least 25 kg to be eligible. Patients must be able to read the consent form and give informed consent. Parent or legal guardians of patients who are minors will sign the informed consent form.
* Patients must have a Karnofsky performance status of at least 80.
* LDH ≤ 2x upper limit of normal value; albumin ≥ 3.5 mg/dl. Creatinine ≤ 2mg/dl and AST ≤ 2- fold upper limit of normal.
* A CBC prior to vaccination with WBC ≥ 3000, platelets ≥ 100,000.
* A negative serum bHCG within 2 weeks of vaccination in women of childbearing age.
* Patients must be free of detectable brain metastases. (Brain MRI or CT pre-protocol)

Exclusion Criteria:

* Patients may not be receiving or have received chemotherapy, immunotherapy or radiation therapy within the previous 4 weeks or nitrosourea chemotherapy within the previous 6 weeks. Patients must be fully recovered from any previous therapy or surgery.
* Patients may not have been previously immunized with vaccines containing tyrosinase or gp100, or peptides derived from tyrosinase or gp100.
* Creatinine > 2mg/dl (or history of Creatinine > 2 mg/dl) and AST ≥ 2 fold upper limit of normal.
* Any medical condition or use of medication (e.g., active autoimmune disease, immunodeficiency or corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to respond immunologically to vaccines is grounds for exclusion, at the discretion of the Principal Investigator or co-Principal Investigators. Patients may not have taken systemic corticosteroids (orally or intravenously) within the previous 6 weeks. Inhaled or nasal steroids are permitted.
* Patients who have preexisting retinal or choroidal eye disease (except as outlined in section 5.1.1) will be excluded.
* Patients with serious underlying medical conditions, active infections requiring antimicrobial drugs, or active bleeding will be ineligible.
* Pregnant women, women who are less than 3 months post-partum or women who are nursing are not eligible. Women of childbearing age and sexually active men must be using appropriate contraception during the course of this study and for 3 months following completion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To establish the safety and a recommended dose of subcutaneous human GM-CSF DNA given in conjunction with a multi-epitope peptide vaccine in patients with AJCC stage IIB, IIC, III and IV melanoma who are HLA-A2+. | Up to 15 years post treatment,
To evaluate serum pharmacokinetics of GM-CSF after subcutaneous administration of human GM-CSF DNA. | All patients entered in the Dose Ranging study will undergo pharmacokinetic studies during their first course of therapy.
If toxicities are encountered in the dose ranging part of the study, to establish the maximum tolerated dose (MTD) and dose limiting toxicities (DLT). | If toxicities less than DLT are encountered, then patients will continue on the study at the assigned dose level.
In the immunological efficacy study, to evaluate the immunogenicity of a multi-epitope peptide vaccine. | Up to 15 years post treatment.

SECONDARY OUTCOMES:
A secondary endpoint is to observe the patients for evidence of any anti-tumor response that is generated after vaccination. | Up to 15 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel-Angel Perales, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm